CLINICAL TRIAL: NCT01282450
Title: Concurrent and Non-concurrent Chemo-radiotherapy or Radiotherapy Alone for Patients With Oligo-metastatic Stage IV Non-small Cell Lung Cancer (NSCLC).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: MAASTRO clinic, MAASTRO clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Oligometa's
Record Dates: First submitted 2010-12-06; First posted 2011-01-25 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Stage IV (Oligo-metastases); Non-small Cell Lung Cancer
Keywords: Radiotherapy; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Surgical Procedures, Operative; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Eligible patients
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy
  Other Names: Radiotherapy with or without surgery or chemotherapy

SUMMARY:
In recent years, it has become clear, that also in non-small cell lung cancer (NSCLC), a group of patients with less than 5 distant metastases may experience long-term survival when treated radically to all macroscopic cancer sites. Thus has mostly been established for individuals with so-called solitary brain metastases and to a lesser extend in solitary adrenal gland metastases, but in other metastatic subgroups, the same may be applicable. In a prospective survey in the region of the Integral Cancercentre (IKL), we could identify on a yearly base 30 patients with NSCLC who could theoretically be amendable for radical treatment of all oligo-metastatic locations. We therefore want to perform a prospective study in which patients with less than 4 oligo-metastatic sites from a primary NSCLC will be treated radically with the aim to improve long-term survival. As many discussion points remain, even after thorough discussions with chest physicians, pulmonary surgeons and colleagues from diagnostic disciplines, we decided to go for a pragmatic approach, implying that all macroscopic disease sites should be treated radically, being defined as surgery with a R0 resection or in case of an unforeseen R1 resection, followed by radiotherapy, or radiotherapy to a biological equivalent of at least 60 Gy in 30 daily fractions. In the same patient, one metastatic site may be treated with surgery and another with radical radiotherapy. Systemic treatment was not made mandatory, because it was felt that it's role is unclear in patients with early stage local cancer and with oligo-metastatic disease.

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radical radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes to an MLD (Mean Lung Dose) of 20 +/- 1Gy, irrespective of lung function and/or to all metastatic sites to a minimal biological equivalent of 60Gy in 30 daily fractions. This may be delivered with hypofractionated stereotactic techniques or with other more protracted fractionation regimen.

Both the primary tumor, the regional N1 lymph nodes and the oligo-metastatic site(s) may be treated with surgery, as long as an R0 resection is deemed possible. Systemic treatment is not required, but should be given according to the local extend of the tumor.

Local radiotherapy will be delivered according to the protocol of MAASTRO clinic for that anatomical site.

Other dose-constraints: spinal cord max: 54Gy, brachial plexus (Dmax): 66Gy The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven NSCLC
* UICC stage IV, or solitary metastases (< 5), which are amendable for radical local treatment
* Performance status 0-2
* Other malignancy is allowed if controlled at the point of diagnosis

Exclusion Criteria:

* Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
* Stage I-III, except for T4 because of pleural metastases
* Performance status 3 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  The survival of participating patient two years after entering the study
Overall survival | 3 years
  The survival of participating patients, three years after entering the study.

SECONDARY OUTCOMES:
Progression free survival | 2 years
Dyspnea (CTC4.0) | 2 years
Dysphagia (CTC 4.0) | 2 years
Patterns of recurrence | 2 years
Progression free survival | 3 years
Dyspnea (CTC4.0) | 3 years
Dysphagia (CTC4.0) | 3 years
Patterns of recurrence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — MAASTRO clinic, Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] De Ruysscher D, Wanders R, van Baardwijk A, Dingemans AM, Reymen B, Houben R, Bootsma G, Pitz C, van Eijsden L, Geraedts W, Baumert BG, Lambin P. Radical treatment of non-small-cell lung cancer patients with synchronous oligometastases: long-term results of a prospective phase II trial (Nct01282450). J Thorac Oncol. 2012 Oct;7(10):1547-55. doi: 10.1097/JTO.0b013e318262caf6. PMID 22982655